CLINICAL TRIAL: NCT03756324
Title: The Effect of Chinese Herbal Medicine for Reducing the Application of Antibiotics in the Treatment of Acute Mastitis With Three Groups in Randomized Controlled Trial.
Brief Title: The Effect of Chinese Herbal Medicine for Reducing the Application of Antibiotics in the Treatment of Acute Mastitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Collaborators: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaohua Pei, Principal Investigator, Clinical Professor, Academic Leader of Breast Disease in Traditional Chinese Medicine., Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFH2018-7032
Record Dates: First submitted 2018-11-18; First posted 2018-11-28 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Mastitis Acute Female
Keywords: Pugongying; Herba Taraxaci; Acute Mastitis; Cefdinir; Randomized controlled trial; Postpartum; Breastfeeding; Lactation; multicenter; Chinese herb; Traditional Chinese medicine; Cephalosporin; Antibiotics
MeSH Terms: conditions — Breast Feeding | interventions — Cefdinir; Educational Status; Medical Order Entry Systems

STUDY DESIGN:
Intervention Model Description: Based on previous studies, considering the 20% expulsion rate, the investigators plan to recruit 306 participants with sample-size calculation formula. The sequence of randomization (1:1:1) will be generated by the statisticians with a computer program.
Who Masked: Outcomes Assessor
Masking Description: Due to the different numbers of interventions, the investigators can not blind the participants and the doctors. Thus, the CRF recorders, outcomes assessors and the statisticians will be blinded in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHPM (Chinese Herbal Patent Medicine ) (Experimental): CHPM (Chinese Herbal Patent Medicine ): Pugongying (Herba Taraxaci) Granules, 15g/tid for 3 days, follow-up for 7 days.
  Education, basic medical order.
  Interventions: Drug: CHPM (Chinese Herbal Patent Medicine ); Behavioral: Education
- CHPM & Antibiotics Cefdinir Capsules (Experimental): CHPM (Chinese Herbal Patent Medicine): Pugongying (Herba Taraxaci) granules, 15g/tid for 3 days, follow-up for 7 days.
  Antibiotics: Cefdinir Capsules, 0.1g/tid for 2 days, follow-up for 7 days.
  Education, basic medical order.
  Interventions: Drug: CHPM (Chinese Herbal Patent Medicine ); Behavioral: Education; Drug: Antibiotics Cefdinir Capsules
- Antibiotics Cefdinir Capsules (Active Comparator): Antibiotics: Cefdinir Capsules, 0.1g/tid for 3 days, follow-up for 7 days.
  Education, basic medical order.
  Interventions: Drug: Antibiotics Cefdinir Capsules; Behavioral: Education

INTERVENTIONS:
Drug: CHPM (Chinese Herbal Patent Medicine ) — Pugongying (Herba Taraxaci) granules is named as Pugongying Granules in China and produced by Kunming pharmaceutical factory co. LTD. The form is granules, and the participants will take the medicine after dissolved as 15g/tid for 3 days, and the investigators will follow them up for 7 days when the participants are stopped administrating.
  Other Names: Pugongying (Herba Taraxaci) Granules
  Arms: CHPM & Antibiotics Cefdinir Capsules; CHPM (Chinese Herbal Patent Medicine )
Drug: Antibiotics Cefdinir Capsules — Cefdinir Capsules is also named as Cefdinir and produced by Astellas Pharma Inc. The form is capsule, and participants will take orally the capsules with water as 0.1g/tid for 3 days, and the investigators will follow them up for 7 days when the participants are stopped administrating.
  Other Names: Cefdinir Capsules of "normal course group"
  Arms: Antibiotics Cefdinir Capsules
Behavioral: Education — Doctors will give suggestions and the medical orders to all participants, including dietary, emotional regulation and the knowledge of breast-feeding.
  Other Names: Basic medical order; Medical order
Drug: Antibiotics Cefdinir Capsules — Cefdinir Capsules is also named as Cefdinir and produced by Astellas Pharma Inc. The form is capsule, and participants will take orally the capsules with water as 0.1g/tid for 2 days, and the investigators will follow them up for 7 days when the participants are stopped administrating.
  Other Names: Cefdinir Capsules of "short course group"
  Arms: CHPM & Antibiotics Cefdinir Capsules

SUMMARY:
The object of the study is to evaluate the effect of Pugongying (Herba Taraxaci) Granules to reduce the application of antibiotics for women with acute mastitis.

DETAILED DESCRIPTION:
Acute mastitis affects the health and quality of life of the infants and mothers during the lactation. Increasing studies indicate that bacterial infections and/or dysbacteriosis are essential to the mechanisms of the disease. Thus, antibiotics is widely used in clinical practice, especially cephalosporin in China. However, mistaking antibiotic will affect the physical function, even mothers' breastfeeding. The previous clinical trial that the investigators had conducted in the Third affiliated hospital of Beijing University of Chinese Medicine, has demonstrated that Chinese herbal medicine can act better than Cefdinir in the fever-relief time and breast pain scores. Some studies the investigators searched in the databases have showed that Pugongying (Herba Taraxaci) has a broad spectrum of antimicrobial activity, and it can regulate dysbacteriosis. At the same time, Pugongying (Herba Taraxaci) can also promote the secretion of milk and maintain the patency of milk well. The main ingredient of Pugongying (Herba Taraxaci) Granules is Pugongying herbs (Herba Taraxaci). Pugongying (Herba Taraxaci) Granules is approved by China Food and Drug Administration (CFDA) to treat acute mastitis. Although Pugongying (Herba Taraxaci) Granules is widely used in clinical practice, there is no trial to test the efficacy of Pugongying (Herba Taraxaci) for women with acute mastitis. Therefore, the investigators set three groups with Pugongying (Herba Taraxaci) Granules alone, Cefdinir alone and combination of Pugongying (Herba Taraxaci) Granules and Cefdinir.

ELIGIBILITY:
Inclusion Criteria:

1. Women in lactation who have strong willing to breastfeeding;
2. The course of acute mastitis should be within 3 days, and the ultrasound examination indicates there is no abscess cavity formed;
3. The body temperature is higher than 37.2°C but lower than 41°C;
4. The VAS scores of participants≥4;
5. Patients with acute mastitis have not received other medical therapies;
6. Those who have signed informed consent.

Exclusion Criteria:

1. Participants who suffered nipple ulceration, painful fissuring or developmental defects fail to breastfeed;
2. Participants with other breast diseases are not appropriate to breastfeed;
3. Participants with severe cognitive or metabolic diseases will affect breastfeeding;
4. Participants who have been allergic to penicillin and cephalosporin.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of fever-relief | Measured from the beginning to the end of the treatment, every 4 hours for 3 days, total 19 times including the baseline measured, specifically on 2:00 am, 6:00 am, 10:00 am, 14:00 pm, 18:00 pm, 22:00 pm.
  Body temperature will be measured by mercury thermometer and recorded on the prepared card by participants. The temperature of the participants reduces to 37.2℃ or more below, assessing as the normal temperature. And the normal temperature last for at least 24 hours, considered as fever-relief.
  To evaluate the effect of drug action time and the temperature changing from the baseline to the end of 3-day treatment.
Change of the sores of breast pain | Measured from the beginning to the end of the treatment, every 8 hours for 3 days, total 10 times including the baseline measured, specifically measured on 6:00 am, 14:00 pm, 22:00 pm.
  Pain of breast will be self-reported by participants and recorded. A visual analog scale (VAS) is used to assess breast pain. The scale was tested in the investigator's previous trial. 0 score indicates "no uncomfortable feeling". 1-3 indicates "mild uncomfortable feeling". 4-6 indicates "moderate uncomfortable feeling". 7-10 indicates "severe uncomfortable feeling".
  To evaluate the changing from the baseline to the end of 3-day treatment.
Change of the area of the breast masses | The masses will be measured from the beginning to the end of the treatment, once a day for 3 days, and recorded with a camera, total 4 times including the baseline measured.
  The masses are manual outlined by the outcome assessor.
  To evaluate the changing from the baseline to the end of 3-day treatment.

SECONDARY OUTCOMES:
The patency of milk | The outcome will be measured from the beginning to the end of the treatment, once a day for 3 days, total 4 times including the baseline measured.
  The 0-3 scores are used to describe the patency of milk from no stagnation to severe stagnation. 0 indicates that there is no stagnation with breast and milk spurts out by slightly pressure; 1 indicates mild stagnation and milk flows by more pressure; 2 indicates moderate stagnation and milk drops out by much more pressure; 3 indicates there is severe stagnation and no milk excreted. The outcome will be measured by the outcome assessor.
  To evaluate the changing from the baseline to the end of 3-day treatment.
The scores of Traditional Chinese Medicine (TCM) symptoms | Measured from the beginning to the end of the treatment, once a day for 3 days, total 4 times including the baseline measured.
  The assessment criteria refer to Standard of diagnosis and treatment in TCM symptoms (2016 version, released by State Administration of Traditional Chinese Medicine of the People's Republic of China). The outcome is specifically used to assess the holistic physical status of the participants and will be measured by TCM practitioners.
  To evaluate the changing from the baseline to the end of 3-day treatment.
Change of the White blood cell count | Routine blood test will be tested and analyzed by laboratory at the beginning since enrolling and after 3-day treatment.
  Measured by the routine blood test.
  To evaluate the changing from the baseline to the end of 3-day treatment.
Change of the percentage of neutrophil | Routine blood test will be tested and analyzed by laboratory at the beginning since enrolling and after 3-day treatment.
  Measured by the routine blood test.
  To evaluate the changing from the baseline to the end of 3-day treatment.
Change of the C-reactive protein. | Routine blood test will be tested and analyzed by laboratory at the beginning since enrolling and after 3-day treatment.
  Measured by the routine blood test.
  To evaluate the changing from the baseline to the end of 3-day treatment.
Number of participants with treatment-related adverse events | Symptoms of allergic reaction will be observed at any time. Signs examination will be taken once a day, for 3 days, total 4 times including the baseline measured. Laboratory test will be taken at the beginning since enrolling and after 3-day treatment.
  Adverse events are assessed by CTCAE (version 5.0, released by NIH and NIC). The outcomes measured at baseline are used to determine whether the participants are eligible to participate the study and the outcomes measured during and after 3-day treatment are used to assess the safety of the intervention medicine and to protect the rights of the participants.
  To focus on (1) allergic reaction; (2) the vital signs: resting heart rate in times/minutes, respiratory rate in times/minutes and blood pressure in mmHg; (3) laboratory test: urinalysis (LEU, BLO, KET, NIH, GLU, PRO, UBG, SG) in positive/negative, stool routine (Sed occult blood) in postive/negative, electrocardiogram in normal/abnormal, liver function test (AST, ALT, TBIL, DBIL, TG, GLU) in positive/negative and renal function test (CR, UA, UREA) in positive/negative.
  To observe the incidence of the adverse events.

OTHER OUTCOMES:
The incidence of acute mastitis relapse in 3-day follow-up | After 3-day treatment, the participants will be called each day to answer the questions from the investigators, lasting for 3 days.
  After 3-day treatment, the participants will be followed up for 3 days to figure out the incidence of acute mastitis relapse. The investigators will call the participants to inquiry their conditions (body temperature, breast pain, amount of milk).
The indidence of surgery | Clinical evaluation will be conducted after 3-day treatment.
  After 3-day treatment, clinical evaluation will be conducted by doctors. If B-ultrasound shows there is mammary abscess, the doctor will perform surgery based on liquefaction and size of the abscess.
The quantity of additional intervention medicine administration | Clinical evaluation will be conducted after 3-day treatment.
  After 3-day treatment, clinical evaluation will be conducted by doctors. If B-ultrasound shows there is mammary abscess, the doctor will prescribe Cefdinir or Pugongying granules based on liquefaction and size of the abscess.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Pei, MD, Principal Investigator — Beijing University of Chinese Medicine
Locations (3):
- China (3):
  - Beijing Hospital of Traditional Chinese Medicine, Beijing
  - Beijing University of Chinese Medicine Third Affiliated Hospital, Beijing
  - Tongzhou Maternal & Child Health Hospital of Beijing, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin X, Xiao J, Lu C, Ma W, Fan Y, Xue X, Xia Y, Chen N, Liu J, Pei X. Breastmilk microbiome changes associated with lactational mastitis and treatment with dandelion extract. Front Microbiol. 2023 Nov 13;14:1247868. doi: 10.3389/fmicb.2023.1247868. eCollection 2023. PMID 38029215